CLINICAL TRIAL: NCT02709824
Title: Efficacy of an Anti-Discoloration System (ADS) to Reduce Dental Staining in a 0.12% Chlorhexidine-based Mouthwash
Brief Title: Anti-staining Efficacy of Anti-Discoloration System (ADS) Added to Chlorhexidine (CHX)
Acronym: CHX+ADS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Responsible Party: Principal Investigator, ANDREA SARDELLA, Associate Professor, University of Milan
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: ADS2012
Record Dates: First submitted 2016-03-11; First posted 2016-03-16 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Adverse Effect
MeSH Terms: interventions — chlorhexidine gluconate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chlorhexidine gluconate with ADS (Active Comparator): Chlorhexidine 0.12% plus Anti-Discoloration System Mouthwash
  Interventions: Drug: Chlorhexidine gluconate with ADS
- Chlorhexidine gluconate without ADS (Active Comparator): Chlorhexidine 0.12% Mouthwash
  Interventions: Drug: Chlorhexidine gluconate without ADS

INTERVENTIONS:
Drug: Chlorhexidine gluconate with ADS — Oral rinsing, twice a day, for 21 days
  Other Names: Curasept (0.12% Chlorhexidine gluconate with ADS)
  Arms: Chlorhexidine gluconate with ADS
Drug: Chlorhexidine gluconate without ADS — Oral rinsing, twice a day, for 21 days
  Other Names: Dentosan (0.12% Chlorhexidine gluconate without ADS)
  Arms: Chlorhexidine gluconate without ADS

SUMMARY:
Dental staining is the most common local side effect of chlorhexidine (CHX) mouthwashes.

A prospective, cross-over, randomized clinical trial will be carried out in triple blind to compare the effect on dental staining of two 0.12% CHX mouthwashes: with or without anti-discoloration system (ADS). Twenty-two healthy subjects will be enrolled. Briefly, the study includes two sequential stages: in the first phase, the "immediate" objective and subjective evaluation of dental discoloration by spectroscopic and questionnaire-based analyses will be recorded, at baselines and after each 21-days-long cycle of mouthwash. A wash-out period between the cycles of 21 days will be performed.

In the second phase, a long-term (after 6 months) subjective evaluation of dental discoloration will be obtained by means of clinical photograph visual analysis and new questionnaires.

DETAILED DESCRIPTION:
In the first phase, the "immediate" objective and subjective evaluation of dental discoloration by spectroscopic (CIE L*a*b* data analysis with DeltaE evaluation) and questionnaire-based analyses will be recorded. Immediate visual analysis of tooth pigmentation will be evaluated by volunteer him/herself, using a mirror, and by a single dentist soon after the end of each treatment. Participants will indicate the presence/absence of dental pigmentation, and to quantify it with a numeric scale (0= no pigmentation to 10= very strong pigmentation).

These analyses will be performed at baselines and after each 21-days-long cycle of mouthwash.

A wash-out period between the cycles of 21 days will be performed. In the second "late" phase, a long-term subjective evaluation of dental discoloration will be obtained by means of the visual analysis of clinical photograph and new questionnaires. After 6 months from clinical trial (second stage of the study), frontal dental images of volunteers, collected during the first phase, will be printed on photographic paper and, then, visually analyzed, in blind, by the 22 volunteers themselves, as well as by 14 dentists and 13 oral hygienists ad hoc recruited. Dentists and oral hygienists, in particular, will be asked to observe two images of all the 22 subjects, i.e. after treatment with A or B mouthwash, and to answer to the question: "Which picture shows the most pigmented teeth?" Possible answers will be: "A, or B or no difference between the two images". Pigmentation will be also quantified using the numeric scale (0= no pigmentation to 10=strong pigmentation).

The observer will be not instructed in how the color of the teeth should appear in case of CHX pigmentation.

ELIGIBILITY:
Inclusion Criteria:

* to be free from oral mucosa conditions affecting its integrity
* to avoid drug or mouthwash intake during the study and in the previous month

Exclusion Criteria:

* specific allergy to mouthrinses
* presence of periodontitis
* frequent use of Chlorhexidine-based oral hygiene products

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2011-12; Primary Completion 2012-02 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Dental Staining - spectroscopic evaluation | 21 days
  dental color before and after the two treatments

SECONDARY OUTCOMES:
Dental Staining - visual evaluation | 21 days
  dental color before and after the two treatments
Dental Staining - visual evaluation on images | 21 days of treatments, re-analysis of images after 6 months from the end of the trial
  dental color before and after the two treatments

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carrassi, MD, Principal Investigator — University of Milan
Locations (1):
- University of Milan, Milan, Italy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cortellini P, Labriola A, Zambelli R, Prato GP, Nieri M, Tonetti MS. Chlorhexidine with an anti discoloration system after periodontal flap surgery: a cross-over, randomized, triple-blind clinical trial. J Clin Periodontol. 2008 Jul;35(7):614-20. doi: 10.1111/j.1600-051X.2008.01238.x. Epub 2008 Apr 16. PMID 18422695
- [Background] Bernardi F, Pincelli MR, Carloni S, Gatto MR, Montebugnoli L. Chlorhexidine with an Anti Discoloration System. A comparative study. Int J Dent Hyg. 2004 Aug;2(3):122-6. doi: 10.1111/j.1601-5037.2004.00083.x. PMID 16451475
- [Background] Solis C, Santos A, Nart J, Violant D. 0.2% chlorhexidine mouthwash with an antidiscoloration system versus 0.2% chlorhexidine mouthwash: a prospective clinical comparative study. J Periodontol. 2011 Jan;82(1):80-5. doi: 10.1902/jop.2010.100289. Epub 2010 Jul 27. PMID 20653433
- [Background] Li W, Wang RE, Finger M, Lang NP. Evaluation of the antigingivitis effect of a chlorhexidine mouthwash with or without an antidiscoloration system compared to placebo during experimental gingivitis. J Investig Clin Dent. 2014 Feb;5(1):15-22. doi: 10.1111/jicd.12050. Epub 2013 Jun 14. PMID 23766285